CLINICAL TRIAL: NCT05385471
Title: A Phase Ia Clinical Trial to Assess the Safety and Immunogenicity of the Blood-stage Malaria Candidate Vaccines RH5.1 in Matrix-M and R78C in Matrix-M, Both Alone and in Combination, in Healthy UK Adults
Brief Title: A Phase Ia Clinical Trial to Assess the Safety and Immunogenicity of the Blood-stage Malaria Candidate Vaccines RH5.1 in Matrix-M and R78C in Matrix-M in Healthy UK Adults
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC089
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Malaria, Falciparum
Keywords: R78C; RH5.1; Matrix-M
MeSH Terms: conditions — Malaria, Falciparum | interventions — Matrix-M

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): 8+1 volunteers receiving three doses of 10 µg R78C with 50 µg of Matrix-M on days 0, 28 and 182 via intramuscular (IM) injection in the deltoid region of the non-dominant arm
  Interventions: Biological: Matrix M with R78C and/or RH5.1
- Group 2 (Experimental): 8+1 volunteers receiving three doses of 10 µg R78C + 10 µg RH5.1 with 50 µg of Matrix-M on days 0, 28 and 182 via intramuscular (IM) injection in the deltoid region of the non-dominant arm
  Interventions: Biological: Matrix M with R78C and/or RH5.1
- Group 3 (Experimental): 8+1 volunteers receiving three doses of 10 µg RH5.1 with 50 µg of Matrix-M on days 0, 28 and 56 via intramuscular (IM) injection in the deltoid region of the non-dominant arm
  Interventions: Biological: Matrix M with R78C and/or RH5.1
- Group 4 (Experimental): 8+1 volunteers receiving two doses of 10 µg R78C + 10 µg RH5.1 with 50 µg of Matrix-M on days 0, 28, one dose of 10 µg R78C with 50 µg of Matrix-M on day 182 and one dose of 10 µg RH5.1 with 50 µg of Matrix-M on day 210, all administered via intramuscular (IM) injection in the deltoid region of the non-dominant arm
  Interventions: Biological: Matrix M with R78C and/or RH5.1

INTERVENTIONS:
Biological: Matrix M with R78C and/or RH5.1 — 50 µg of Matrix-M adjuvant with R78C and/or RH5.1 at different doses and timepoints

SUMMARY:
This is an open-label, single-centre Phase I P. falciparum blood-stage vaccine trial to assess the safety and immunogenicity and efficacy of the candidate malaria vaccines R78C and RH5.1 formulated in adjuvant Matrix-M

DETAILED DESCRIPTION:
Volunteers will be recruited into one of four groups (n=8+1 per group) at the Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford. Volunteers in groups 1, 2 and 4 will be followed up for a total of approximately 12 months. There will be 3 sentinel participants in each group (and for each successive vaccination), which will require an independent safety review prior to each successive vaccination. Group 3 is not a first-in-human group and so can be recruited at any time and participants will be followed up for a total of approximately 20 months from first vaccination. All volunteers will be given 10 µg R78C and/or 10 µg RH5.1 soluble protein in combination with 50 µg of Matrix-M via intramuscular (IM) injection in the deltoid region of the non-dominant arm.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adult aged 18 to 45 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their GP
* Participants of childbearing potential only: must practice continuous effective contraception until 3 months after the final study vaccination (see section 9.10)
* Agreement to refrain from blood donation for the duration of the study
* Able and willing to provide written informed consent to participate in the trial

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* History of clinical malaria (any species) or previous participation in any malaria vaccine trial or controlled human malaria infection trial
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months
* Use of immunoglobulins or blood products (e.g. blood transfusion) in the last three months
* Receipt of any vaccine in the 30 days preceding enrolment, or planned receipt of any other vaccine within 30 days following each study vaccination, with the exception of COVID-19 vaccines, which should not be received between 14 days before to 7 days after any study vaccination
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period
* Concurrent involvement in another clinical trial involving an investigational product or planned involvement during the study period
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data, as assessed by the Investigator
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of anaphylaxis in reaction to vaccinations
* Pregnancy, lactation or intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition that may affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol misuse as defined by an alcohol intake of greater than 25 standard UK units every week
* Suspected or known injecting drug use in the 5 years preceding enrolment
* Hepatitis B surface antigen (HBsAg) detected in serum
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless volunteer has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV ribonucleic acid (RNA) PCR at screening for this study)
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of R78C in Matrix-M™ and RH5.1 in Matrix-M in healthy adult volunteers at alone and in combination by assessing the occurrence of solicited local reactogenicity signs and symptoms for 7 days following each vaccination | 7 days following each vaccination
  Occurrence of solicited local reactogenicity signs and symptoms for 7 days following each vaccination. These will be tabulated, detailing frequency, duration and severity of AEs. Haematological and biochemical laboratory values will be presented according to local grading scales.
To assess the safety of R78C in Matrix-M™ and RH5.1 in Matrix-M in healthy adult volunteers at alone and in combination by assessing the occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following each vaccination | 7 days following each vaccination
  Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following each vaccination. These will be tabulated, detailing frequency, duration and severity of AEs. Haematological and biochemical laboratory values will be presented according to local grading scales.
To assess the safety of R78C in Matrix-M™ and RH5.1 in Matrix-M in healthy adult volunteers at alone and in combination by assessing the occurrence of unsolicited adverse events for 28 days following the vaccination | 28 days following the vaccination
  Occurrence of unsolicited adverse events for 28 days following the vaccination. These will be tabulated, detailing frequency, duration and severity of AEs. Haematological and biochemical laboratory values will be presented according to local grading scales.
To assess the safety of R78C in Matrix-M™ and RH5.1 in Matrix-M in healthy adult volunteers at alone and in combination, assessed through the number of participants with abnormal laboratory test results | 28 days following vaccination
  Occurrence of change from baseline laboratory tests
To assess the safety of R78C in Matrix-M™ and RH5.1 in Matrix-M in healthy adult volunteers at alone and in combination, assessed through the number of participants with serious adverse events | Whole duration of the Study (up to day 600 depending on group)
  Occurrence of serious adverse events during the whole study duration. Haematological and biochemical laboratory values will be presented according to local grading scales.

SECONDARY OUTCOMES:
To assess the humoral immunogenicity of R78C in Matrix-M™ and RH5.1 in Matrix-M when administered to healthy volunteers alone and in combination assessing antigen-specific IgG antibody levels, with comparison before and after vaccination | From a number of key timepoints, baseline up to day 600 (dependant on group)
  Serum ELISA response, quantitative antigen-specific IgG antibody levels (µg/mL readout) over time - analysis of peak responses and longevity, with comparison before and after vaccination
To assess the humoral immunogenicity of R78C in Matrix-M™ and RH5.1 in Matrix-M in healthy volunteers assessing antigen-specific antibody subclass/isotype measurement, with comparison before and after vaccination | From a number of key timepoints, baseline up to day 600 (dependant on group)
  Serum ELISA response, antigen-specific antibody subclass/isotype measurement, with comparison before and after vaccination
To assess the humoral immunogenicity of R78C in Matrix-M™ and RH5.1 in Matrix-M in healthy volunteers assessing antigen-specific antibody avidity measurement, with comparison before and after vaccination | From a number of key timepoints, baseline up to day 600 (dependant on group)
  Serum ELISA response, antigen-specific antibody avidity measurement, with comparison before and after vaccination
To assess the humoral immunogenicity of R78C in Matrix-M™ and RH5.1 in Matrix-M when administered to healthy volunteers alone and in combination assessing In vitro GIA, with comparison before and after vaccination | From a number of key timepoints, baseline up to day 600 (dependant on group)
  In vitro GIA against 3D7 clone P. falciparum parasites using purified total IgG and a single-cycle pLDH readout assay, with comparison before and after vaccination
To assess the humoral immunogenicity of R78C in Matrix-M™ and RH5.1 in Matrix-M in healthy volunteers assessing Purified IgG ELISA versus GIA titration "Quality Analysis", with comparison before and after vaccination | From a number of key timepoints, baseline up to day 600 (dependant on group)
  Purified IgG ELISA versus GIA titration "Quality Analysis"

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Minassian, DPhil FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom